CLINICAL TRIAL: NCT06308315
Title: Effects of Rhythmic Balance Auditory Vision Training And Strength Training On Motor Function And Cognition In Children With Autism Spectrum Disorder.
Brief Title: Effects of Rhythmic Balance Auditory Vision Training And Strength Training With Autism Spectrum Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0297
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Cognition; Motor function; Strength training
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient would be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Rhythmic Training+ Routine Physical therapy) (Experimental): Rhythmic balance auditory vision training will be given thrice a week for 8 weeks. it is a 45 minute training program that consist of:
  1. 5 minute warm up activities (arm swings).
  2. Bal-A-Vis-X training thrice a week for 20 minutes.
  3. 5-minute cool down activities.
  Routine Physical therapy treatment for 15 minutes
  Interventions: Other: Rhythmic balance visual auditory exercise + Routine physical therapy
- Group B (Strength Training+ Routine Physical Therapy) (Experimental): Strength training Program will be performed thrice a week for 8 weeks. session of 45 minute will be given to the patient. The expert managed sessions based on:
  10-min warm-up activities, 25-min basic exercise 10- min cool-down activities.
  Interventions: Other: Strength Training + Routine Physical Therapy

INTERVENTIONS:
Other: Rhythmic balance visual auditory exercise + Routine physical therapy — 5 minute warm-up activities.
  Bal-A-Vis-X training includes:
  1. Ball Rectangle; A and B hold one ball in each hand, simultaneously bounce right balls to patient left hand; while balls bounce, clap left balls on right hand; catch patient ball with left hand; continue pattern. Bounces must be simultaneous. (10 minutes)
  2. Ball rectangle in which one hand has to toss a ball to a partner and the other hand catch an incoming bag from the partner and 2 ball drop/pass/catch, two-foot jumping forward, tandem walking on ground. (10 minutes)
  Routine Physical therapy treatment includes:
  Range of Motion exercises, Stretching, Strength, balance training for 15 minutes
  5 minute cool-down activities.
  Arms: Group A (Rhythmic Training+ Routine Physical therapy)
Other: Strength Training + Routine Physical Therapy — The expert managed sessions based on:
  5 minute warm-up activities. 5 minute cool-down activities. Strength training includes 5 tasks for 20 minutes
  1. core strengthening,
  2. upper and lower limbs strength in both static positions as well as with dynamic movements
  3. standing long jump,
  4. knee push-ups,
  5. sit-ups
  Routine Physical therapy treatment will be given for 15 minutes.
  It includes:
  Range of Motion exercises, Stretching, Strength, balance training.
  Arms: Group B (Strength Training+ Routine Physical Therapy)

SUMMARY:
Autism, a complex neurodevelopmental disorder that is marked by limited interests, and challenges in communication and social interactions and problem includes difficulties in understanding and responding to social cues, repetitive behaviors, intense focus on specific interests, and challenges with verbal and nonverbal communication. Rhythmic Balance Auditory Vision Training (RBAVT) a therapeutic approach which helps in improving coordination and balance in individuals with various neurological conditions. Strength training enhance physical health and muscle development. Thus, the purpose of this study is to compare the effects of rhythmic balance auditory vision training and strength training on motor function and cognition in children with autism spectrum disorder.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted in Autism center Lahore. Sample of 76 patients will be recruited in this trial by using the convenience sampling technique. Participants will be randomly allocated in two groups using lottery method. Group A will receive Rhythmic balance visual auditory exercise. Group B will receive strength training exercises. Both groups will receive routine physical therapy as baseline treatment. All the participants will receive 3 sessions per week for 12 weeks.Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) will be used assessment tool to measure fine and gross motor skills and Wisconsin Card Sorting Test (WCST) will be assessment tool that evaluates cognitive flexibility and problem-solving abilities.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 6 and 12 years.
2. Rating Scale (CARS) with scores ranging from 30 to 36.
3. Confirmation of the diagnosis of autism by a psychiatrist based on Diagnostic and Statistical manual of Mental Disorders.
4. Physical and cognitive ability

Exclusion Criteria:

1. Children with history of auditory, visual, or respiratory deficits, or fixed deformities of the extremities.
2. Medical contraindications such as orthopedic or acute conditions that hinder participation in the exercise program.
3. History of psychotropic medication within the last 4 weeks.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) | 12th week
  The Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) is a widely used assessment tool to measure fine and gross motor skills in individuals aged 4 to 20. It evaluates various aspects of motor proficiency, including running speed, balance, coordination, and fine motor control. The test helps identify motor skill strengths and weaknesses to aid in intervention and treatment planning. The BOTMP test is a valid assessment tool with 8 subscales (53 sections) for evaluating motor functions. The shortened version has 8 subscales (14 sections), assessing gross motor skills (4 subscales), fine motor skills (3 subscales), and a subscale evaluating both. Its test-retest reliability stands at 87%.

SECONDARY OUTCOMES:
Wisconsin Card Sorting Test (WCST) | 12th week
  The Wisconsin Card Sorting Test (WCST) is a psychological assessment tool that evaluates cognitive flexibility and problem-solving abilities. The WCST includes 4 stimulus cards and 128 response Cards. One red triangle, 2 green stars, 3 yellow crosses, or 4 blue circles are demonstrated in the stimulus cards. The 128 response cards contain pictures combining different shapes (triangles, stars, crosses, & circles), colors (red, blue, yellow, & green), and numbers (1, 2, 3, or 4). The cards are presented on a screen in the computer Version of the WCST. The participant has to choose an Answer card for matching with one of the 4 key cards Based on its potential characteristics with 4 cards. The reliability estimates for the accurate sorts, categories, and perseverative errors were within the favorable range (rel ≥ .90)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD-PT, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No